CLINICAL TRIAL: NCT06937060
Title: Effect of Semaglutide in Patients With Psoriasis and Obesity
Acronym: SEMPSO
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Chung Man Ho Martin, Honorary Clinical Assistant Professor, The University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UW 25-083
Record Dates: First submitted 2025-04-15; First posted 2025-04-20 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-04

CONDITIONS: Psoriasis (PsO); Obesity and Overweight
Keywords: semaglutide; obesity; psoriasis
MeSH Terms: conditions — Psoriasis; Obesity; Overweight | interventions — semaglutide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Active (alternative intervention) (Experimental): Semaglutide is act as an adjunct to a reduced calorie diet and increase physical activity for chronic weight management in obesity or overweighted adult. Initiate Semaglutide with a dosage of 0.25 mg injected subcutaneously once-weekly, from week 1 to week 24, i.e. 24 dosage of Semaglutide in total.
  Interventions: Biological: semaglutide

INTERVENTIONS:
Biological: semaglutide — Semaglutide is act as an adjunct to a reduced calorie diet and increase physical activity for chronic weight management in adult with an initial body mass index (BMI) of 30 kg/m2 or greater (obesity) or 27 kg/m2 or greater (overweight) in the presence of at least one weight-related comorbid condition (e.g., hypertension, type 2 diabetes mellitus, or dyslipidemia)

SUMMARY:
Obesity is well known to be an important comorbidity of psoriasis. It gives rise to higher risk of psoriatic arthritis, more severe disease and also poorer response to biologics. Weight loss can lead to reduction in psoriasis severity. Previous studies had demonstrated the efficacy of older glucagon-like peptide-1 receptor agonist (GLP1 RA) on improvement of psoriatic disease activity. Effective weight loss has been achieved by newer GLP1 RA.7 It is also known to reduce cardiovascular outcomes in patient without diabetes. Trials on the effect of semaglutide on psoriasis has not been performed except case reports.

Semaglutide is an injectable prescription medicine that may help adults and children aged 12 years and older with obesity or some adults with excess weight (overweight) who also have weight-related medical problem to help them lose weight. It contains a GLP1 RA indicated as an adjunct to diet and exercise to improve glycemic control. It has potential anti-inflammatory effects on top of weight reduction, that may lead to improvement in psoriatic disease activity.

This is an open-label, single-armed, prospective pilot trial on obese, psoriasis patients. The investigators aim to recruit 14 patients. Patients will be maintained on standard care for their psoriasis. Add-on treatment with semaglutide of up to 2.0mg per week will be administered to the intervention arm in addition to lifestyle intervention. Treatment with previous systemic immunosuppressants is allowed.

The maximum study duration for a single subject in the study will be approximately 36 weeks, 4 weeks of screening, 24-week treatment period, and a 12-week safety follow up period after the last study dose of semaglutide at week 24.

ELIGIBILITY:
Inclusion Criteria:

* a clinical diagnosed Psoriatic disease of at least 6 months before signing of informed consent.
* Women who are sexually active and not postmenopausal, agreement to remain abstinent or use 2 effective methods of contraception
* >18 years of age, up to 75 years of age
* Adult with an initial body mass index (BMI) of 30 kg/m2 or greater (obesity) or 27 kg/m2 or greater (overweight) in the presence of at least one weight-related comorbid condition (e.g., hypertension, type 2 diabetes mellitus, or dyslipidemia)
* Moderate to severe psoriasis (PASI score 5-10= moderate, >10 = severe)
* Chinese ethnicity
* On stable dose of standard treatment
* Ability to comply with stud

Exclusion Criteria:

* Patients who refuse to give consent
* Contraindication to use of GLP1 RA
* History of pancreatitis
* History of MEN / MTC
* Known hypersensitivity to semaglutide or excipients in semaglutide
* Type 1 diabetes
* Gallbladder disease
* Active malignancy or History of malignancy within 5 years
* Active chronic or acute infection requiring treatment with systemic antibiotics, antiviral, antiparasitic, antiprotozoal, or antifungals within 4 weeks before baseline visit
* Pregnancy or breastfeeding, subjects should inform their healthcare provider of a known or suspected pregnancy
* History of allergic reaction assessed as related to investigational product by the investigator
* Major psychiatric illness
* Treatment with live/ attenuated vaccine within the last 28 days prior to randomisation
* History of alcohol or substance abuse within 6 months prior to initial screening
* Patients with a history of suicidal attempts or active suicidal ideation

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2025-03-20 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2027-01-31 (Estimated)

PRIMARY OUTCOMES:
Change in mean Psoriasis Area and Severity Index (PASI) before and after semaglutide treatment. | 36 weeks
  The change in mean Psoriasis Area and Severity Index (PASI) score before and after semaglutide treatment will be assessed. The PASI score is a widely used tool to measure the severity and extent of psoriasis. It combines the assessment of the severity of lesions (erythema, induration, and desquamation) and the area affected into a single score. The PASI score ranges from 0 to 72, where 0 indicates no disease and 72 represents the most severe disease.

CONTACTS AND LOCATIONS:
Overall Officials: Man Ho Martin Chung, Principal Investigator — The University of Hong Kong
Locations (1):
- The University of Hong Kong, Department of Medicine, Hong Kong, Hong Kong